CLINICAL TRIAL: NCT01347593
Title: Prophylactic Ceftizoxime (Cefizox) for Elective Cesarean Delivery in Soba Hospital Sudan
Brief Title: Prophylactic Ceftizoxime (Cefizox) for Elective Cesarean Delivery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Khartoum (Other)
Collaborators: Ministry of Health, Sudan (Unknown)
Responsible Party: Principal Investigator, Ishag Adam, Professor, University of Khartoum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ceftizoxime cesarean
Record Dates: First submitted 2011-05-02; First posted 2011-05-04 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Caesarean
Keywords: ceftizoxime; Cesarean; post caesarean febrile morbidity
MeSH Terms: interventions — Ceftizoxime

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ceftizoxime (cefizox) injection (Experimental): ceftizoxime (cefizox) as single dose of 1 g at the interval of 30-60 minutes before the incision
  Interventions: Drug: ceftizoxime

INTERVENTIONS:
Drug: ceftizoxime — ceftizoxime (cefizox) injection either after clamping the cord
  Other Names: cefizox

SUMMARY:
Ceftizoxime (Cefizox) will reduce post Cesarean delivery febrile morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Elective Cesarean section

Exclusion Criteria:

* Diabetes severe anaemia allergy

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 220 (Actual)
Dates: Start 2011-05; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
reducing post Cesarean section febrile morbidity | 4 days
  reducing infection rate

CONTACTS AND LOCATIONS:
Locations (1):
- Soba Hospital, Khartoum, Khartoum State, Sudan

REFERENCES:
- [Derived] Osman B, Abbas A, Ahmed MA, Abubaker MS, Adam I. Prophylactic ceftizoxime for elective cesarean delivery at Soba Hospital, Sudan. BMC Res Notes. 2013 Feb 8;6:57. doi: 10.1186/1756-0500-6-57. PMID 23394621